CLINICAL TRIAL: NCT02655224
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-385 40 mg in the Treatment of Pain Symptoms Associated With Uterine Fibroids
Brief Title: A Placebo-Controlled, Phase 3 Study of Relugolix (TAK-385) 40 mg in the Treatment of Pain Symptoms Associated With Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-385-3008; U1111-1178-1086 (Registry Identifier: WHO); JapicCTI-163127 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Uterine Fibroids
Keywords: Drug Therapy
MeSH Terms: conditions — Leiomyoma | interventions — relugolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relugolix 40 mg (Experimental): Relugolix placebo-matching tablet, orally, once daily before breakfast for 3 to 6 weeks in the run-in period, followed by relugolix 40 mg, tablet, orally once daily before breakfast for 12 weeks.
  Interventions: Drug: Relugolix
- Placebo (Placebo Comparator): Relugolix placebo-matching tablet, orally, once daily before breakfast for 3 to 6 weeks in the run-in period, followed by relugolix placebo-matching tablet, orally once daily before breakfast for 12 weeks.
  Interventions: Drug: Relugolix placebo

INTERVENTIONS:
Drug: Relugolix — Relugolix Tablets
  Other Names: TAK-385
  Arms: Relugolix 40 mg
Drug: Relugolix placebo — Relugolix placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Relugolix (TAK-385) in patients having pain symptoms associated with uterine fibroids.

DETAILED DESCRIPTION:
The drug being tested in this study is called relugolix (TAK-385). Relugolix is being tested to treat people who have uterine fibroids.

The study enrolled 65 patients. Participants received relugolix placebo in run in period for 3 to 6 weeks. After run-in period, participants were randomly assigned to one of the two treatment groups in 1:1 ratio:

1. Relugolix 40 mg
2. Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants were asked to take one tablet at the same time each day throughout the study.

This multi-center trial was conducted in Japan. The overall time to participate in this study was 20 to 28 weeks, including run-in period of 3 to 6 weeks and a treatment period of 12 weeks. Participants made multiple visits to the clinic, and 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Entering the Screening Period (at VISIT 1)

1. In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. Prior to VISIT 1, the participant has a diagnosis of uterine fibroids confirmed by transvaginal ultrasound, abdominal ultrasound, magnetic resonance imaging (MRI), computed tomography (CT), or laparoscopy, and has never received any surgical treatment for the myoma (measurable noncalcified myoma with a longest diameter of ≥3 cm).
4. The participant is a premenopausal Japanese woman.
5. The participant is aged 20 years or older on the day of signing and dating the informed consent form.
6. The participant has 1 or more measurable noncalcified myomas with a longest diameter of ≥3 cm confirmed by transvaginal ultrasound.
7. The participant has experienced 1 or more regular menstrual cycles (25 to 38 days) immediately prior to VISIT 1 and that should include menstrual bleeding for at least 3 consecutive days.
8. The participant who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the study.

   Inclusion Criteria for Entering the Run-in Period (at VISIT 2)
9. The participant has experienced regular menstrual cycles (25 to 38 days) immediately prior to VISIT 2 that should include menstrual bleeding for at least 3 consecutive days (at least 2 regular menstruation cycles to be confirmed by Inclusion criteria #7 and #9).

   Inclusion Criteria for Entering the Treatment Period (at VISIT 3)
10. The participant has 1 or more measurable noncalcified myomas, with a longest diameter of ≥3 cm confirmed by transvaginal ultrasound (the same myoma should be measured in Inclusion criterion #6).
11. The participant has a maximum Numerical Rating Scale (NRS) score of ≥4 during 1 menstrual cycle just before VISIT 3.
12. The participant has pain symptoms associated with uterine fibroids for at least 2 days during 1 menstrual cycle just before VISIT 3.
13. The participant has experienced regular menstrual cycles (25 to 38 days) after VISIT 1 that should include menstrual bleeding for at least 3 consecutive days (at least 3 regular menstruation cycles to be confirmed by Inclusion criteria #7, #9 and #13).

Exclusion Criteria:

1. The participant has received any investigational compound within 24 weeks prior to the start of the administration of the study drug for the day of first menstruation after VISIT 1.
2. The participant has received relugolix (including placebo) in a previous clinical study.
3. The participant is an immediate family member or study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, or sibling) or may consent under duress.
4. The participant has lower abdominal pain due to irritable bowel syndrome or severe interstitial cystitis.
5. The participant has a current history of thyroid gland disorder with irregular menstruation, or has a potential for irregular menstruation due to thyroid gland disorder, as determined by the investigator or subinvestigator.
6. The participant has a previous or current history of pelvic inflammatory disease within 8 weeks prior to VISIT 1.
7. The participant has a positive Pap smear test result obtained within 1 year prior to VISIT 1 (if there are no previous test results, those who were judged positive in the test conducted before VISIT 2).
8. The participant has a history of panhysterectomy or bilateral oophorectomy.
9. The participant has had markedly abnormal uterine bleeding or anovulatory bleeding, as determined by the investigator or subinvestigator.
10. The participant has a malignant tumor or a history of a malignant tumor within 5 years prior to VISIT 1.
11. The participant has been treated with selective estrogen receptor modulators (SERMs) (excluding drugs for external use and dietary supplements) within 4 weeks prior to VISIT 2.
12. The participant has been treated with any of the following drugs within 8 weeks prior to VISIT 2: oral contraceptive or sex hormone preparations (norethindrone, norethisterone, medroxyprogesterone, estrogen, or other progestins), and within 16 weeks prior to VISIT 2: gonadotropin-releasing hormone (GnRH) analogues, dienogest, danazol, or aromatase inhibitors (for 1- and 3-month sustained-release preparations, within 20 and 28 weeks prior to VISIT 2, respectively).
13. The participant has a previous or current history of severe hypersensitivity or severe allergies to drugs.
14. The participant has nondiagnosable abnormal genital bleeding.
15. Female participant who is pregnant, lactating, or intending to become pregnant or to donate ova prior to the signing of informed consent, during the study period, or within 1 month after the end of the study.
16. The participant has clinically significant cardiovascular disease (eg, myocardial infarction or unstable angina pectoris within 24 weeks prior to VISIT 1) or uncontrollable hypertension (eg, resting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg at Screening and Run-in Period).
17. The participant is ineligible for this study based on standard 12-lead electrocardiogram (ECG) findings, as determined by the investigator or subinvestigator.
18. The participant has active liver disease or jaundice, or with alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin (total bilirubin) >1.5 times the upper limit of normal (ULN) in the clinical laboratory tests at VISIT 1 and 2.
19. The participant has a previous or current history of diseases considered to be ineligible for this study, including severe hepatic impairment, jaundice, renal impairment, cardiovascular disease, endocrine system disease, metabolic disorder, pulmonary disease, gastrointestinal disease, neurological disease, urological disease, immune disease, mental disorder (especially depression-like symptoms) and suicide attempt resulting from a mental disorder.
20. The participant has a previous or current history of drug abuse (defined as any illicit drug use) or alcohol abuse.
21. The participant is ineligible for this study for other reasons, as determined by the investigator or subinvestigator.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-03-26 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- Japan (11):
  - Matsudo, Chiba
  - Ebetsu, Hokkaido
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Ibaraki, Osaka
  - Sakai, Osaka
  - Bunkyo-ku, Tokyo
  - Minato-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Kagoshima
  - Osaka

REFERENCES:
- [Derived] Osuga Y, Enya K, Kudou K, Hoshiai H. Relugolix, a novel oral gonadotropin-releasing hormone antagonist, in the treatment of pain symptoms associated with uterine fibroids: a randomized, placebo-controlled, phase 3 study in Japanese women. Fertil Steril. 2019 Nov;112(5):922-929.e2. doi: 10.1016/j.fertnstert.2019.07.013. Epub 2019 Oct 6. PMID 31594635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 15 investigative sites in Japan from 26 March 2016 to 19 May 2017.
Pre-assignment Details: Participants with a diagnosis of uterine fibroids were enrolled in a 1:1 ratio in one of two treatment groups: relugolix 40 mg or placebo.
Period: Overall Study
Arm/Group | Relugolix 40 mg | Placebo
Started | 33 | 32
Completed (Completed=Completed Treatment) | 32 | 31
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relugolix 40 mg | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (3.95) | 42.6 (5.24) | 41.5 (4.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 33 | 32 | 65
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 157.5 (6.40) | 159.2 (4.25) | 158.3 (5.48)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 57.55 (11.775) | 57.47 (11.511) | 57.51 (11.555)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body Mass Index = weight (kg)/[height (m)^2]
  kilogram per square meter (kg/m^2) | 23.15 (4.146) | 22.56 (3.714) | 22.86 (3.919)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 20 | 21 | 41
  Current Smoker | 6 | 8 | 14
  Ex-Smoker | 7 | 3 | 10
Birth Experience [Count of Participants; unit: Participants]
  Had Birth Experience | 12 | 12 | 24
  Had No Birth Experience | 21 | 20 | 41
Type of Uterine Fibroid [Count of Participants; unit: Participants]
  Subserosal Fibroid | 17 | 9 | 26
  Intramural Fibroid | 22 | 29 | 51
Stopped Any Medications for Uterine Fibroids [Count of Participants; unit: Participants]
  Had Stopped Any Medications | 5 | 7 | 12
  Had not Stopped Any Medications | 28 | 25 | 53
Number of Participants With No Surgery for Uterine Fibroids [Count of Participants; unit: Participants] | 33 | 32 | 65
Volume of Myoma [Mean (Standard Deviation); unit: cm^3] | 78.83 (84.189) | 101.38 (172.738) | 89.94 (134.633)
Volume of Uterus [Mean (Standard Deviation); unit: cm^3] | 252.29 (202.938) | 300.09 (295.341) | 275.82 (251.837)
Maximum Numerical Rating Scale (NRS) Score [Mean (Standard Deviation); unit: score on a scale] — Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain.
  score on a scale | 6.64 (1.817) | 6.28 (1.689) | 6.46 (1.751)
Uterine Fibroid Symptom and Quality of Life (UFS-QOL) Score: Symptom Severity [Mean (Standard Deviation); unit: score on a scale] — UFS-QOL was a 37-item self-reporting tool for evaluating QOL in participants with uterine fibroid. It includes eight symptom-related questions and 29 HRQL questions across six subscales (concern, activities, energy/mood, control, self-consciousness, sexual function). The total symptom severity score is ranging from 0 to 100. The higher scores indicate greater severity.
  score on a scale | 25.5 (8.59) | 30.3 (13.07) | 27.9 (11.20)
UFS-QOL Score: Health Relate Quality of Life (HRQL) Total [Mean (Standard Deviation); unit: score on a scale] — UFS-QOL was a 37-item self-reporting tool for evaluating QOL in participants with uterine fibroid. It includes eight symptom-related questions and 29 HRQL questions across six subscales (concern, activities, energy/mood, control, self-consciousness, sexual function). The total HRQL score is ranging from 0 to 100. The higher scores indicate better QOL.
  score on a scale | 83.9 (12.47) | 80.0 (15.00) | 82.0 (13.81)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Maximum NRS Score of 1 or Less During the 28 Days Before the Final Dose of Study Drug
Description: Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain. The percentage of participants with a score of 1 or less is reported.
Time Frame: For 28 days before the final dose of study drug (up to Week 12)
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study drug for the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
percentage of participants | 57.6 | 3.1
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Test type: Superiority — The point estimate and 2-sided 95% confidence interval of odds ratio were calculated between relugolix 40 mg group and placebo group; p < 0.0001, Fisher's Exact Test; Odds Ratio (OR) = 42.071, 95% CI 2-sided [5.113 to 346.181] — Relugolix 40 mg/Placebo

2. Secondary Outcome: Percentage of Participants With a Maximum NRS Score of 0 During the 28 Days Before the Final Dose of Study Drug
Description: Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain. The percentage of participants with a score of 0 is reported.
Time Frame: For 28 days before the final dose of study drug (up to Week 12)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug for the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
percentage of participants | 48.5 | 3.1
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 29.176, 95% CI 2-sided [3.555 to 239.478] — Relugolix 40 mg/Placebo

3. Secondary Outcome: Mean NRS Score During the 28 Days Before the Final Dose of Study Drug
Description: Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain.
Time Frame: For 28 days before the final dose of study drug (up to Week 12)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
score on a scale | 0.50 (0.967) | 0.99 (1.274)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Test type: Other — The mean differences between relugolix 40 mg group and placebo group and the two-sided 95% confidence intervals were calculated; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.050 to 0.069] — Relugolix 40 mg-Placebo

4. Secondary Outcome: Percentage of Days Without Pain Symptoms (NRS = 0) During the 28 Days Before the Final Dose of Study Drug
Description: Percentage of day without pain symptoms (NRS = 0) was reported. Number of days without pain symptoms is determined by a zero score on the NRS. Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain. Percentage of days without pain symptoms (NRS=0) during the 28 days before the final dose of study drug (%) = [(number of days without pain symptoms (NRS=0) during the last 28 days of the treatment)/(number of days with available data during the last 28 days of the treatment)]*100.
Time Frame: For 28 days before the final dose of study drug (up to Week 12)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
percentage of days | 76.73 (32.006) | 64.78 (29.015)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 11.96, 95% CI 2-sided [-3.201 to 27.112] — Relugolix 40 mg-Placebo

5. Secondary Outcome: Percentage of Participants With Maximum NRS Score of 1 or Less From Day 1 to 28, From Day 29 to 56, and From Day 57 to 84
Description: as for outcome 1
Time Frame: Day 1 to 28, Day 29 to 56, and Day 57 to 84
Population: FAS included all participants who were randomized and received at least 1 dose of study drug for the treatment period. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
percentage of participants
  Day 1 to 28 | 24.2 | 0.0
  Day 29 to 56: number analyzed (Participants) | 33 | 31
  Day 29 to 56 | 45.5 | 12.9
  Day 57 to 84: number analyzed (Participants) | 32 | 31
  Day 57 to 84 | 59.4 | 12.9
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Day 29 to 56; Test type: Other — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.625, 95% CI 2-sided [1.605 to 19.709] — Relugolix 40 mg/Placebo. Statistical analysis for Day 29 to 56 and Day 57 to 84, the odds ratio was calculated. For Day 1 to 28, its ratio was not calculated due to zero cell
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Placebo; Day 57 to 84; Test type: Other — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 9.865, 95% CI 2-sided [2.784 to 34.955] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants With a Maximum NRS Score of 0 From Day 1 to 28, From Day 29 to 56, and From Day 57 to 84
Description: as for outcome 2
Time Frame: Day 1 to 28, Day 29 to 56, and Day 57 to 84
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
percentage of participants
  Day 1 to 28 | 15.2 | 0.0
  Day 29 to 56: number analyzed (Participants) | 33 | 31
  Day 29 to 56 | 27.3 | 6.5
  Day 57 to 84: number analyzed (Participants) | 32 | 31
  Day 57 to 84 | 46.9 | 6.5
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Day 29 to 56; Test type: Other — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.438, 95% CI 2-sided [1.071 to 27.609] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Placebo; Day 57 to 84; Test type: Other — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 12.794, 95% CI 2-sided [2.603 to 62.880] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Mean NRS Score From Day 1 to 28, From Day 29 to 56, and From Day 57 to 84
Description: as for outcome 3
Time Frame: Day 1 to 28, Day 29 to 56, and Day 57 to 84
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
score on a scale
  Day 1 to 28 | 1.26 (1.490) | 1.17 (1.141)
  Day 29 to 56: number analyzed (Participants) | 33 | 31
  Day 29 to 56 | 0.59 (0.991) | 1.16 (1.457)
  Day 57 to 84: number analyzed (Participants) | 32 | 31
  Day 57 to 84 | 0.43 (0.776) | 0.97 (1.279)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Day 1 to 28; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Each Period) = 0.09, 95% CI 2-sided [-0.574 to 0.745] — Relugolix 40 mg-Placebo
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Placebo; Day 29 to 56; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Each Period) = -0.57, 95% CI 2-sided [-1.190 to 0.049] — Relugolix 40 mg-Placebo
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Placebo; Day 57 to 84; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Each Period) = -0.54, 95% CI 2-sided [-1.074 to -0.012] — Relugolix 40 mg-Placebo

8. Secondary Outcome: Percentage of Days Without Pain Symptoms (NRS = 0) From Day 1 to 28, From Day 29 to 56, and From Day 57 to 84
Description: Percentage of day without pain symptoms (NRS = 0) was reported. Number of days without pain symptoms is determined by a zero score on the NRS. Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain. Percentage of days without pain symptoms (NRS=0) (%) = [(number of days without pain symptoms (NRS=0) during the last 28 days of the treatment)/(number of days with available data during the last 28 days of the treatment)]*100.
Time Frame: Day 1 to 28, Day 29 to 56, and Day 57 to 84
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
percentage of days
  Day 1 to 28 | 60.49 (34.043) | 56.32 (28.891)
  Day 29 to 56: number analyzed (Participants) | 33 | 31
  Day 29 to 56 | 73.98 (31.718) | 61.29 (31.459)
  Day 57 to 84: number analyzed (Participants) | 32 | 31
  Day 57 to 84 | 77.43 (30.854) | 65.84 (29.224)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Placebo; Day 1 to 28; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Each Period) = 4.17, 95% CI 2-sided [-11.507 to 19.839] — Relugolix 40 mg-Placebo
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Placebo; Day 29 to 56; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Each Period) = 12.70, 95% CI 2-sided [-3.098 to 28.494] — Relugolix 40 mg-Placebo
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Placebo; Day 57 to 84; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Each Period) = 11.60, 95% CI 2-sided [-3.554 to 26.745] — Relugolix 40 mg-Placebo

9. Secondary Outcome: Number of Participants Reporting Who Had One or More Treatment-emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to Week 16
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 29 | 18

10. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Vital Signs
Description: Vital signs included sitting blood pressure (after the participant has rested for at least 5 minutes), body temperature (oral or tympanic measurement) (degree Celsius [°C]) and pulse (beats per minute [bpm]) are reported.
Time Frame: Up to Week 16
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
Participants
  Diastolic Blood Pressure Lower (<50 mmHg) | 2 | 1
  Body temperature Lower (<35.6 °C) | 4 | 2

11. Secondary Outcome: Number of Participants With TEAEs Related to Weight
Description: Number of participants with TEAEs of which threshold was 5% or above in either treatment group related to weight was reported.
Time Frame: Up to Week 16
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With TEAEs Related to Standard 12-lead Electrocardiogram (ECG)
Description: Number of participants with TEAEs of which threshold was 5% or above in either treatment group related to ECG was reported.
Time Frame: Up to Week 16
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Laboratory Tests
Description: Number of participants with any markedly abnormal values in laboratory tests collected throughout study is reported. WBC = White blood cells, GGT = gamma-glutamyl transferase, LLN = lower limit of normal or lower reference limit, ULN = upper limit of normal or upper reference limit.
Time Frame: Up to Week 16
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Placebo
Number analyzed (Participants) | 33 | 32
Participants
  Hemoglobin Lower (<0.8×LLN g/dL) | 0 | 1
  WBC Upper (>1.5×ULN × 10^3cells/μL) | 0 | 1
  Total Cholesterol Upper (>300 mg/dL) | 2 | 0
  Triglycerides Upper (>2.5×ULN mg/dL) | 0 | 3
  Total Bilirubin Upper (>2.0 mg/dL) | 1 | 0
  GGT Upper (>3×ULN U/L) | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 16
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Relugolix 40 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 27/33 | 14/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix 40 mg (N=33) | Placebo (N=32)
Viral upper respiratory tract infection (Infections and infestations) | 7 | 9
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Headache (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 0
Metrorrhagia (Reproductive system and breast disorders) | 13 | 3
Menorrhagia (Reproductive system and breast disorders) | 4 | 3
Menstruation irregular (Reproductive system and breast disorders) | 1 | 3
Genital haemorrhage (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 0
Hot flush (Vascular disorders) | 15 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT02655224/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02655224/SAP_001.pdf